CLINICAL TRIAL: NCT03621124
Title: Maladaptive Adipose Tissue Activity in Cancer
Status: Terminated | Type: Observational
Why Stopped: COVID-19 Pandemic
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-17-13470; NCI-2018-01510 (Other: NCI CTRP); P30CA016059 (NIH); HM20009089 (Other: IRB No.)
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cancer Nos
MeSH Terms: conditions — Neoplasms | interventions — Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brown Adipose Tissue Positive patients: Patients with known malignancy and incidental finding of positron emission tomography/ computerized tomography (PET/CT) scans positive for brown adipose tissue (BAT). After obtaining informed consent and all initial screening visit procedures, patients will participate in two four-hour recording sessions in the whole room indirect calorimeter to assess resting energy expenditure, and patient's thermal (comfort) response to the temperature of the room.
  Interventions: Procedure: Resting Energy Expenditure; Other: Thermal Comfort Questionnaire
- Brown Adipose Tissue Negative Patients: Patients with known malignancy and no evidence of brown adipose tissue BAT activity positron emission tomography/ computerized tomography (PET/CT) scans to be matched to group 1 for primary tumor and stage, sex, age (±5 years), BMI (±3 Kg/m2). After obtaining informed consent and all initial screening visit procedures, patients will participate in two four-hour recording sessions in the whole room indirect calorimeter to assess resting energy expenditure, and patient's thermal (comfort) response to the temperature of the room.
  Interventions: Procedure: Resting Energy Expenditure; Other: Thermal Comfort Questionnaire

INTERVENTIONS:
Procedure: Resting Energy Expenditure — During each visit, the participant will be assessed in a resting state in a stable temperature controlled environment, and will undergo tests to find out how the body adjusts its metabolism to different temperatures.
  Other Names: ENRGEXP
Other: Thermal Comfort Questionnaire — Patients will be given a questionnaire to assess their thermal response (whether they felt warmer or colder) during each study visit.

SUMMARY:
The purpose of this pilot research is to study brown adipose tissue, a type of fat that increases metabolism (burns energy) during exposure to cold, and how it may contribute to the weight loss observed in cancer.

DETAILED DESCRIPTION:
The purpose of this research is to study brown adipose tissue, a type of fat that increases metabolism (burns energy) during exposure to cold, and how it may contribute to the weight loss observed in cancer. Many patients affected by cancer lose weight, despite normal or increased nutrition. It may progress to the condition called "cancer-associated cachexia." Cancer associated cachexia is defined by an ongoing loss of skeletal muscle mass with or without the loss of fat mass, and may negatively affect quality of life and the ability to undergo cancer treatments. Metabolism is the breakdown of food by the body into the energy that your body needs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 years of age
* Have active cancer diagnosis.
* Have had a PET/CT scan within the past 12 months at time of enrollment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current use of beta-blockers
* Women who are pregnant or unsure of their pregnancy status
* Women who are breastfeeding
* Suffers from severe claustrophobia
* Diagnosed with a serious psychiatric condition which could impede the judgement of the investigators, and/or the successful conduct of the recording.
* In remission stage for cancer diagnosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients equal to or greater than forty years of age with an active cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Difference in resting energy expenditure between brown adipose tissue (BAT)-positive and BAT-negative patients with cancer. | 27 Months
  Characterization of the energy metabolism profiles of cancer patients with and without evidence of BAT activation will be assessed utilizing one sided t-test.

SECONDARY OUTCOMES:
Difference in energy expenditure between room temperature and response to warm exposure (energy expenditure) in BAT-positive and BAT-negative cancer patients. | 27 Months
  Assessment of environmental modulation as an effective strategy to mitigate maladaptive BAT activation in patients with malignancy will be assessed by two-sided t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco S Celi, MD, MHSc, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/ Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No